CLINICAL TRIAL: NCT00003683
Title: Treatment of Sarcomatous Kidney Cancer That is Metastatic in Adults With Doxorubicin and Ifosfamide. Phase II Study
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066785; FRE-FNCLCC-REINSARDI; EU-98057
Record Dates: First submitted 1999-11-01; First posted 2004-01-27 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Doxorubicin; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: doxorubicin hydrochloride
Drug: ifosfamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining doxorubicin and ifosfamide in treating patients who have metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy in terms of objective response after treatment with ifosfamide and doxorubicin in patients with metastatic sarcomatoid renal cell cancer. II. Determine the toxicity of this regimen in these patients. III. Determine the effect of this regimen on the survival of these patients.

OUTLINE: This is a multicenter study. Patients receive doxorubicin IV on day 1 and ifosfamide IV over 2 hours on days 1 and 2. Treatment is repeated every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic, sarcomatoid renal cell carcinoma Measurable disease At least 15 mm for pulmonary sites At least 20 mm for other sites No uncontrolled CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: Greater than 3 months Hematopoietic: Neutrophil count greater than 1500/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 9 g/dL Hepatic: Bilirubin less than 1.5 times normal Transaminases less than 2 times normal (less than 4 times normal if due to liver metastases) Renal: Creatinine less than 1.6 mg/dL Creatinine clearance greater than 60 mL/min Other: No contraindication to anthracycline treatment No unstable major organ defect No prior malignancy except basal cell skin cancer or carcinoma in situ of the uterus Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1998-03 (Actual); Primary Completion 2000-11-05 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Culine, MD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (14):
- France (14):
  - Institut Sainte Catherine, Avignon
  - Centre Leon Berard, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - C.H.U. - Hopital Gaston Doumergue, Nîmes
  - Hotel Dieu de Paris, Paris
  - Institut Curie - Section Medicale, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Hospitalier General de Saint Nazaire, Saint-Nazaire
  - Institut Gustave Roussy, Villejuif